CLINICAL TRIAL: NCT01922323
Title: Metabolomics of Liver Regeneration Following Partial Hepatectomy in Healthy Living Liver Donors
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 013-140
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Liver Insufficiency
Keywords: Living liver donor
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Each subject will provide samples of urine and blood at specific timepoints as outlined in the protocol
Oversight: Data Monitoring Committee: No

SUMMARY:
The PI will study metabolism during liver regeneration in living liver donors

DETAILED DESCRIPTION:
Samples of blood and urine will be collected from study participants at defined timepoints. The samples will be evaluated to study the metabolism of the regenerating liver after a portion of the liver has been donated from a living donor.

ELIGIBILITY:
Inclusion Criteria:

1. Potential donor must be in excellent medical and psychological health.
2. Potential donor must be between the ages of 18 and 60.
3. Must have a compatible blood type to the recipient.
4. Must have health care coverage for non-donor related health issues that arise post donation
5. Recipient and donor must have compatible body size.
6. Donors Body Mass Index (BMI) must be less than 30.
7. All previous donor abdominal surgeries will be reviewed on a case by case basis by the surgeon.

Exclusion Criteria:

1. Positive blood test for Human Immunodeficiency Virus, Hepatitis C virus, Hepatitis B virus
2. The size of the donor liver is not large enough to safely resection and still retain enough volume to function normally after the surgery.
3. Liver biopsy show liver cirrhosis or early stages of HCC.

   -

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be comprised of living liver donors.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
Characterized Metabolic Changes during liver regeneration | one year after donation

CONTACTS AND LOCATIONS:
Overall Officials: Giuliano Testa, MD, Principal Investigator — Sammons Cancer Center, Baylor University Medical Center
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Bottiglieri T, Wang X, Arning E, Fernandez H, Wall A, McKenna G, Ruiz R, Onaca N, Trotter J, Lawrence M, Naziruddin B, Asrani SK, Testa G. Longitudinal profiling of plasma and urine metabolites during liver regeneration in living liver donors. Clin Transplant. 2022 Jan;36(1):e14490. doi: 10.1111/ctr.14490. Epub 2021 Oct 1. PMID 34545967